CLINICAL TRIAL: NCT02503033
Title: A Phase I, Open-label, Dose-escalation Study of the Safety and Pharmacokinetics of HMPL-523 in Patients With Relapsed or Refractory Hematologic Malignancies
Brief Title: A Study of HMPL-523 in Relapsed or Refractory Hematologic Malignancies
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hutchison Medipharma Limited (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Organization: Hutchmed (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-523-00AU1
Record Dates: First submitted 2015-07-13; First posted 2015-07-20 (Estimated); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Hematologic Malignancies
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HMPL-523 (Experimental): Oral administration, at a dose of 100, 200, 400, 600, 800 and 1000mg once daily or 300mg and 400mg twice daily at Dose-escalation stage.
  At the Dose-expansion stage, HMPL-523 600mg will be dosed once daily.
  Interventions: Drug: HMPL-523

INTERVENTIONS:
Drug: HMPL-523 — Oral administration, once daily

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of HMPL-523 administered to patients with relapsed or refractory Hematologic Malignancies

To determine the maximum tolerated dosage/recommended phase 2 dosage and characterize the dose limited toxicities associated with HMPL-523 when administered to patients with relapsed or refractory Hematologic Malignancies

DETAILED DESCRIPTION:
There are two stages in this study: a dose-escalation stage (stage 1) and a dose-expansion stage (stage 2).

Dose-escalation stage (stage 1). The conventional 3+3 design (3 patients per dose cohort, with the potential to add additional 3 patients to the same cohort to further evaluate toxicity) will be applied for dose escalation and maximum tolerated dosage determination. Approximately 18 to 27 evaluable patients will be enrolled. The actual number of patients depends on the dose limited toxicities situation as well as the maximum tolerated dosage reached at this stage.

Dosing will include QD (quaque die) and bis in die (BID) cohorts. A cycle of study treatment will be defined as 28 days of continuous dosing.

Dose-expansion stage (stage 2). In this stage, approximately 40 patients with B-cell Non-Hodgkin's Lymphomas or Chronic Lymphocytic Leukemia will be enrolled with 600mg once daily as starting dose. The tumor types of the expansion stage are restricted to Chronic lymphocytic leukemia/ small lymphocytic lymphoma (CLL/SLL), Mantle cell lymphoma (MCL), Follicular Lymphoma (FL) (Grade 1-3a), Marginal zone lymphoma (MZL) and Waldenstrom's macroglobulinemia / Lymphoplasmacytic lymphoma (WM/LPL). Subjects will receive HMPL-523 600mg once daily with every 28-day treatment cycle until disease progression, death, or intolerable toxicity, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form.
2. Ability to comply with the protocol.
3. Age>=18 years.
4. ECOG performance status of 0 or 1.
5. Histologically relapsed or refractory chronic lymphocytic leukemia, lymphoma, multiple myeloma(MM) In the dose expansion stage, the tumor types are restricted to relapsed or refractory CLL/SLL, MCL, FL (Grade 1-3a), MZL and WM/LPL.
6. Have failed at least one prior therapy or patients who are unable to tolerate standard therapy or no curative therapy or therapy of higher priority exists.
7. In the dose-expansion stage, patients must have measurable disease for objective response assessment.

   NOTE: measurable disease with FL, MCL, MZL, LPL, or SLL defined as at least 1 bi-dimensionally measurable lesion (>1.5 cm in its largest dimension by computerized tomography [CT] scan)., as defined in appendix 9.
8. Expected survival of more than 24 weeks as determined by the investigator.
9. Male or female patients of child-bearing potential must agree to use double barrier contraception, condoms, sponge, foams, jellies, diaphragm or intrauterine device (IUD), contraceptives (oral or parenteral), Implanon®, injectables or other avoidance of pregnancy measures during the study and for 90 days after the last day of treatment. Post-menopausal females (>45 years old and without menses for >1 year) and surgically sterilized females are exempt from this criterion.

Exclusion Criteria:

1. Patients with primary CNS lymphoma.
2. Known active central nervous system or leptomeningeal lymphoma.
3. Any of the following laboratory abnormalities:

   1. Absolute neutrophil count<1.5×109/L
   2. Hemoglobin <80g/L.
   3. Platelet<75 ×109/L. NOTE: in expansion stage patients with cell counts below the thresholds listed above may be considered eligible if in the investigators opinion the reason is believed to be due to bone marrow infiltration. The investigator will discuss the eligibility of such patients with the sponsor and only upon approval (confirmed in writing) by the sponsor will a patient be enrolled in the study.
4. Inadequate organ function, defined by the following:

   1. Total bilirubin >1.5the ULN with the following exception:

      Patients with known Gilbert disease who have serum bilirubin level ≤3 the ULN and normal AST/ALT may be enrolled.
   2. AST and/or ALT > 2.5 the ULN with the following exception:Patients with documented disease infiltration of the liver may have AST and/or ALT levels ≤ 5 the ULN.
   3. Serum creatinine > 1.5 the ULN or estimated creatinine clearance < 50 mL/min.
   4. Serum amylase or lipase > the ULN.
   5. Triglycerides and/or cholesterol >1.5 the ULN.
   6. International normalized ratio (INR)>1.5 the ULN or activated partial thromboplastin time (aPTT)>1.5 the ULN.

   For patients requiring anticoagulation therapy with warfarin, a stable INR between 2-3 is required. If anticoagulation is required for a prosthetic heart valve, then INR should be between 2.5-3.5 for eligibility NOTE: patients may be considered for the study if liver or kidney function is impaired, but this impairment is believed to be a result of the patient's underlying disease. The investigator will discuss the eligibility of such patients with the Sponsor and only upon approval (confirmed in writing) by the Sponsor will a patient be enrolled in the study.
5. Subjects with presence of clinically detectable second primary malignant tumors at enrollment, or other malignant tumors within the last 2 years (with the exception of radically treated basal cell or squamous cell carcinoma of the skin, in situ cervix, or in situ breast cancer).
6. Any anti-cancer therapy, including chemotherapy, hormonal therapy, biologic therapy, or radiotherapy within 3 weeks prior to initiation of study treatment.
7. Herbal therapy ≤1 week prior to initiation of study treatment.
8. Prior use of any anti-cancer vaccine.
9. Prior treatment with any SYK inhibitors (e.g. Fostamatinib).
10. Prior administration of radioimmunotherapy 3 months prior to initiation of study treatment.
11. Taking strong CYP3A inhibitors, and inducers and drugs metabolized by CYP3A, 2B6 and 1A2 that are identified as narrow therapeutic drugs within 7 days or 3 half-lives, whichever is longer, prior to administration of the first dose of study drug (refer to Appendix 15).
12. Adverse events from prior anti-cancer therapy that have not resolved to Grade ≤1, except for alopecia.
13. Prior autologous transplant within 6 months prior to first dose of study drug.
14. Prior allogeneic stem cell transplant within 6 months prior to initiation of study treatment or with any evidence of active graft versus host disease or requirement for immunosuppressants within 28 days prior to initiation of study treatment.
15. Clinically significant active infection (pneumonia)
16. Major surgical procedure within 4 weeks prior to initiation of study treatment.
17. Clinically significant history of liver disease, including cirrhosis, current alcohol abuse, or current known active infection with HIV, hepatitis B virus (HBV), or hepatitis C virus (HCV).

    Active infection is defined as requiring treatment with antiviral therapy or presence of positive test results for hepatitis B (hepatitis B surface antigen and/or total hepatitis B core antibody) or HCV antibody.

    Patients who test positive for hepatitis B core antibody are eligible only if test results are also positive for hepatitis B surface antibody and polymerase chain reaction (PCR) is negative for HBV DNA.

    Patients who are positive for HCV serology are only eligible if testing for HCV RNA is negative.
18. Pregnant (positive pregnancy test) or lactating women.
19. New York Heart Association (NYHA) Class II or greater congestive heart failure.
20. Congenital long QT syndrome or QTc > 450 msec.
21. Currently use medication known to cause QT prolongation or Torsades de Pointes (http:// www.crediblemeds.org)
22. History of myocardial infarction or unstable angina within 6 months prior to initiation of study treatment.
23. History of stroke or transient ischemic attack within 6 months prior to initiation of study treatment.
24. Inability to take oral medication, prior surgical procedures affecting absorption, or active peptic ulcer disease.
25. Image evidence of gallstone or other bile duct disease within 6 months prior to initiation of study treatment.
26. Treatment within a clinical study within 30 days prior to initiation of study treatment.
27. Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding that, in the investigator's opinion, gives reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or renders the patient at high risk from treatment complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2015-11 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
dose limited toxicities evaluated with NCI CTCAE v4.03 | within 28days after the first dose
  Incidence of dose limited toxicities and associated dose of HMPL-523

SECONDARY OUTCOMES:
maximum plasma concentration calculated with Blood samples | within 29 days after the first dose
  Blood samples will be taken to measure the levels of study drug
time to reach maximum concentration calculated with Blood samples | within 29 days after the first dose
  Blood samples will be taken to measure the levels of study drug
Objective response rate | within 30 days after the last dose
  the proportion of subjects who have a Complete Response or Partial Response
adverse events evaluated by NCI CTCAE v4.03 | from the first dose to within 30days after the last dose
  Incidence of adverse events and associated dose of HMPL-523

CONTACTS AND LOCATIONS:
Overall Officials: Chen Yu, MD, Study Director — Hutchison Medi Pharma
Locations (12):
- Australia (12):
  - Canberra Hospital, Canberra, Australian Capital Territory
  - Border Medical Oncology Research Unit, Albury, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Townsville Hospital, Townsville, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Ballarat Regional Integrated Cancer Centre, Ballarat, Victoria
  - St Vincent's Hospital, Fitzroy, Victoria
  - Peninsula & South Eastern Haematology and Oncology Group, Frankston, Victoria
  - Barwon Health, Geelong, Victoria
  - Austin Hospital, Heidelberg, Victoria
  - Cabrini Health, Melbourne, Victoria
  - Royal Perth Hospital, Perth, Western Australia

IPD SHARING:
Plan to Share IPD: Undecided